CLINICAL TRIAL: NCT03106246
Title: Immune Response to Extracellular Vesicles Released by Human Islets of Langerhans
Brief Title: Circulating Extracellular Vesicles Released by Human Islets of Langerhans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Dr. Steven Paraskevas, Associate Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 15-582-MUHC
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Type1 Diabetes Mellitus; Type2 Diabetes; Islet Cell Transplantation
Keywords: Extracellular vesicles; Autoimmunity; Beta-cell injury
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples. Cellular component will be retained for studies using subject specific peripheral blood mononuclear cells. EV will be purified from plasma and also retained separately.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- New onset T1DM: Newly diagnosed Type I diabetic patients who are hyperglycemic but still C-peptide positive
- T1DM: Patients with established type I diabetes. they are hyperglycemic but C-peptide negative
- T2DM: Patients with established type II diabetes.
- Islet Transplant: Patients who received an islet transplantation for type I diabetes
- Healthy Volunteers: Normoglycemic healthy volunteers

SUMMARY:
Beta-cells release extracellular vesicles (EV) and exosomes under normal and pathophysiologic conditions. These EV contain beta-cell specific autoantigens which may trigger the immune response at the initiation of type 1 diabetes. In this study, beta-cell derived EV will be detected and characterized in human blood samples.

DETAILED DESCRIPTION:
Adult subjects will be recruited with: new onset type 1 diabetes mellitus (T1DM), type 2 diabetes mellitus (T2DM) as well as islet transplant candidates. Blood samples will be collected at defined intervals to determine beta-cell specific EV and determine the utility of this biomarker as a measure of beta-cell stress or injury.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 Diagnosis of type 1 diabetes or type 2 diabetes or islet transplant recipient

Exclusion Criteria:

Unknown diagnosis of diabetes Active infection Immunocompromised Organ transplant recipients not including candidates for islet transplant HIV+ Hepatitis C+ Hepatitis B surface antigen+ Known concurrent malignancy Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed Type I and Type II diabetes, patients undergoing islet transplantation and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Determine the levels of circulating EVs | 2 years
  Based on well-known EV markers, subject plasma samples will be characterized to determine whether these EVs are detectable using small particle flow cytometry.
Determine whether these EVs contain islet-specific antigens | 2 years
  EVs will be further characterized using small particle flow cytometry for known islet-specific antigens such as GAD65 and ZnT8

SECONDARY OUTCOMES:
Mutivariate analysis will be performed with patient parameters and EV parameters | 3 years
  Correlate levels of EVs containing islet specific markers to patient parameters like age, duration of established diabetes, levels of autoantibodies,

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No